CLINICAL TRIAL: NCT05748574
Title: The Sleep Well Observation Study: a Single-arm, Open-label, Prospective Intra-individual Change Controlled, Exploratory Pilot Study
Brief Title: Sleep Well Observation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: A. Vogel AG (Industry)
Collaborators: Daacro GmbH & Co. KG (Unknown); Biochemical Laboratory of the Department of Psychobiology, University of Trier (Unknown); SYNLAB GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5'000'749-1
Record Dates: First submitted 2023-02-20; First posted 2023-02-28 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Sleep Disturbance
Keywords: sleep; herbal supplement; pilot trial
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleep Well Sachet "Treatment" (Experimental): Sachet of Sleep Well direct granulate (2.0 g)
  1 sachet contains: 190 mg standardized dry extract of Melissa officinalis leaf , 75 mg dried pressed juice of fresh Lactuca sativa herb, 0.41 g Magnesiumdicitrate, 0.12 g L-Tryptophan, excipients and natural flavors.
  Interventions: Dietary Supplement: Sleep Well Sachet

INTERVENTIONS:
Dietary Supplement: Sleep Well Sachet — Individuals will take 1 Sleep Well sachet daily over 2 weeks Exception: Two sachets are taken on days 4 and 17 upon acute assessment

SUMMARY:
Insomnia is characterized by the recurring difficulty to fall or remain asleep despite motivation and means to do so. People with insomnia also experience excessive daytime sleepiness and other cognitive impairments while they are awake. Facing the situation mentioned and realizing that especially early preventive measures are needed to fight the increasing costs for treatment of sleep related diseases, effective nutrients might be a good and safe option to improve sleep quality.This single-arm, open-label, prospective, observational exploratory pilot study aims at collecting first data on efficacy and safety of "Sleep Well".

DETAILED DESCRIPTION:
This single-center study is a one-armed, open-label, prospective, observational exploratory pilot study and has a duration of 17 days per participant. A total of 50 healthy participants (n=25 female, n=25 male) aged 18-50 years inclusive reported sleep problems at a preliminary stage to the criteria of the German "S3 guideline non-restorative sleep/sleep disorders - insomnia in adults" for the definition of non-organic insomnia according to ICD-10 (F 51.0) are included into the study.

The total study population of N=50 will include two groups: A subgroup of n=40 will not undergo polysomnographic assessment (nonPSG), a group of n=10 will undergo polysomnographic assessment (PSG), in addition to all other assessments. The nonPSG group has a total of 3 study centre visits (V1, V2, V3) and and the PSG group has two further visits prior to V2 and V3 resulting in five study centre visits (V1, V2-1, V2, V3-1, V3). Except for the PSG, all other assessments are identical in the two groups.

All included individuals will take one Sleep Well sachet daily over an intake period of 14 days with an acute dosage at two visits.

ELIGIBILITY:
Inclusion Criteria:

* • Voluntary, written, informed consent to participate in the study.

  * Male or female aged between 18-50 years (inclusive).
  * Self reported sleep problems precursing the criteria of the German "S3 guideline non-restorative sleep/sleep disorders - insomnia in adults".
  * Habitual bedtime between 9 pm and midnight.
  * Agreement to avoid foods such as pitted fruit, bananas and chocolate 24 hours before saliva sample collection.
  * Willing to download wearable app.
  * Easy access to internet for daily e-diary.
  * Cooling capacities available for storage of saliva samples

Exclusion Criteria:

* • Body mass index (BMI) <18.0 or >30.0 kg/m2.

  * Women who are currently pregnant or breastfeeding.
  * Any known history of a disorder affecting sleep quality, such as narcolepsy, obstructive sleep apnea (OSA), restless leg syndrome (RLS), periodic limb movement syndrome (PLMS) or any organic caused sleep disorders e.g. benign prostatic hyperplasia (BPH), renal insufficiency, hepatopathy, urinary tract infections, irritated bladder, or any psychiatric disorder, e.g. depression, anxiety.
  * Have a significant acute or chronic coexisting illness or any condition which contraindicates entry to the study in the opinion of the Investigator (e.g. migraines, active infections).
  * Previous (last 4 weeks prior to screening) or current intake of drugs that could influence sleep patterns including hormone therapy, health products and oriental herbs.
  * Binge drinking (males >140 g/week, females >70 g/week), heavy smoking (>10 cigarettes/day), high caffeine intake (>10 glasses/day).
  * Self-declared illicit drug use (including cannabis and cocaine) for 3 months prior to screening and during the intervention period.
  * Have a high blood pressure (systolic over 159 mmHg or diastolic over 99 mmHg).
  * Have learning and/or behavioural difficulties such as dyslexia or attention deficit hyperactivity disorder (ADHD).
  * Have a visual impairment that cannot be corrected with glasses or contact lenses (including colour-blindness).
  * History or planned travel to a different time zone within 1 month of the first visit or/and during the study participation.
  * Not fluent in German.
  * Have relevant food allergies/intolerances/sensitivities to any substance in the study product.
  * Have oral disease.
  * Participation in another study with any investigational product within 30 days of screening and during the intervention period.
  * Investigator believes that the participant may be uncooperative and/or noncompliant and should therefore not participate in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2023-06-03 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
Change in perceived sleep quantity/quality | 2 weeks intervention
  Measured as per daily electronic sleep diary entries at home. Comparing pre vs. post intervention assessment.
Change in perceived sleep quantity/quality | 1 day intervention
  Measured as per daily electronic sleep diary entries at home. Comparing pre vs. post intervention assessment.

SECONDARY OUTCOMES:
Change in perceived sleep quantity/quality summarized retrospectively | 2 weeks
  Method: standardized sleep questionnaire SF-B/R. Comparing pre vs. post intervention assessment on site.
Change in daytime sleepiness | 2 weeks
  Pre vs. Post intervention assessment of daytime sleepiness measured with the ESS (Epworth Daytime sleepiness scale) questionnaire
Change in state anxiety | 1 day intervention and 2 weeks
  Pre vs. Post intervention assessment of experienced anxiety symptoms via the STAI-X1 questionnaire
Change in negative emotional state | 2 weeks
  Pre vs. Post intervention assessment of anxiety depression and stress symptoms measured via the DASS-21 questionnaire
Change in quality of life | 2 weeks
  Pre vs. Post intervention assessment of life quality via the WHO-QOL-BREF questionnaire
Change in domain specific cognitive performance | 1 day and 2 weeks
  Pre- vs. Post intervention assessment of domain specific cognitive performance via the COMPASS battery such as attention and vigilance, working memory, spatial memory, memory, executive functions
Change in biomarker for chronic stress | 2 weeks
  Change in biomarker for chronic stress via the salivary evening cortisol level taken at 8 pm on two days pre-intervention and 2 days post intervention
Change in biomarker for sleep readiness | 2 weeks
  Change in biomarker for sleep readiness via the salivary evening melatonin level taken at 8 pm on two days pre intervention and two days post intervention.
Change in biomarker for chronic stress via CAR | 2 weeks
  Change in biomarker for chronic stress via CAR (measured immediately at awakening, +30 min and +45 min thereafter) determined as area under the curve (AUC) and increase in biosamples taken on two days pre intervention and two days post intervention.
Change in PSG-recorded sleep quantity/quality | 1 day intervention and 2 weeks
  Pre vs. Post intervention assessment as measured by the polysomnographic "PSG" assessment using a home portable device
Tolerability of the investigational product in view of subject | 1 day and 2 weeks
  Tolerability of the product as per the self-declaration of the subject - safety assessment
Adverse events | 1 day and 2 weeks
  Frequency and kind of adverse events/medical events during the course of the study - safety assessment
Change in physiological sleep quantity/quality | 1 day and 2 weeks intervention
  Measured by actigraphy (wearable). Comparing pre vs. post intervention assessment as Minutes Asleep (minutes spent in deep, rapid-eye-movement (REM), light or asleep stages), Minutes Awake (number of minutes spent in wake or awake stages), Minutes to fall asleep (number of minutes it took to fall asleep), Time in Bed (number of minutes spent in bed (minutes after wakeup + minutes asleep + minutes awake + minutes to fall asleep))

CONTACTS AND LOCATIONS:
Overall Officials: Juliane Hellhammer, Dr, Principal Investigator — daacro GmbH & Co. KG, Science Park Trier, Max-Planck-Str. 22, 54296 Trier/Germany
Locations (1):
- daacro GmbH & Co. KG, Trier, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No